CLINICAL TRIAL: NCT01530802
Title: Reduction of Intraoperative Blood Loss During Laparoscopic Myomectomy by Temporary Clipping of the Uterine Arteries
Brief Title: Temporary Clipping of the Uterine Arteries During Laparoscopic Myomectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Giuseppe Vercellino, Department of Gynecology, Charité Universitätsmedizin, Berlin - Germany
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: EA4/07906
Record Dates: First submitted 2010-11-01; First posted 2012-02-10 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2010-06

CONDITIONS: Leiomyoma; Laparoscopic Myomectomy
Keywords: laparoscopic myomectomy, leiomyoma, blood loss, uterine artery
MeSH Terms: conditions — Leiomyoma; Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uterine artery clipped (Experimental): Both uterine arteries are temporarily clipped by Yasargil clips during laparoscopic myomectomy.
  Interventions: Procedure: clipping of uterine arteries during laparoscopic myomectomy
- Control group (No Intervention): Conventional laparoscopic myomectomy is performed. (No intervention to temporarily occlude uterine arteries is made)
  Interventions: Procedure: clipping of uterine arteries during laparoscopic myomectomy

INTERVENTIONS:
Procedure: clipping of uterine arteries during laparoscopic myomectomy — For laparoscopy standard instruments were used.For vascular clamping we used titan made YASARGIL vessel clips. The patient is put in a 20° Trendelenburg. The surgeon coagulates a 3-4 cm long segment of peritoneum over the ileopsoas muscle. Along the coagulated segment the peritoneum is opened. The surgeon identifies the ureter at its crossing over the common iliac vessels. After medializing the ureter, the pararectal space is opened and the internal iliac artery is identified and dissected till the origin of the uterine artery. The uterine artery is isolated over a distance of about 2 cm. The vascular clip is placed over the uterine artery. Yasargil Clips are applied exclusively in patients of intervention group. Myomectomy is performed in identical fashion in both groups. At the end of myomectomy the vessel clips are removed. The metroplasty is controlled for hemostasis after reopening of the uterine vessels.

SUMMARY:
The aim is to verify, whether intraoperative temporary clipping of the uterine vessels with vascular clips can reduce blood loss significantly.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for the study when between 18 and 50 years of age,
* diagnosed with either symptomatic or asymptomatic leiomyomata, and with desire to keep the uterus, and whose leiomyomata had a minimal combined diameter of ≥ 4 cm.

Exclusion Criteria:

* patients with severe accompanying medical problems, or
* with psychiatric illnesses, which jeopardize the participation, or
* undergoing treatment affecting coagulation and/or hematopoiesis, and
* patients with suspected malignancy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2007-01; Study Completion 2009-12

PRIMARY OUTCOMES:
Blood loss during laparoscopic myomectomy | perioperative (preop and postoperative day3)
  hemoglobin drop transfusion rate

SECONDARY OUTCOMES:
Patency of uterine artery after laparoscopic clipping | perioperative
  Doppler results of the uterine arteries

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Charite University Hospital, Berlin
  - Bernd Holthaus, Damme